CLINICAL TRIAL: NCT02659865
Title: A Single Ascending Dose Study for the Evaluation of the Effects of LY3039478 on the QT/Corrected QT Interval in Healthy Subjects and Pilot Relative Bioavailability
Brief Title: A Study of LY3039478 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16263; I6F-MC-JJCE (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-01-18; First posted 2016-01-20 (Estimated); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — crenigacestat; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: Placebo (Placebo Comparator): Single oral dose of placebo administered in one of three study periods
  Interventions: Drug: Placebo
- Part A: LY3039478 Capsule Formulation (Formulation 3) (Experimental): Escalating single oral dose of 25 milligram (mg), 50 mg, and 75 mg capsule formulation (formulation 3) LY3039478 administered in two of three study periods
  Interventions: Drug: LY3039478 Capsule Formulation (Formulation 3)
- Part B: LY3039478 Drug-In Capsule (Reference, Formulation 1) (Experimental): Single oral 50 mg dose of drug-in capsule (reference, formulation 1) LY3039478 administered in one of two study periods
  Interventions: Drug: LY3039478 Drug-in Capsule (Reference, Formulation 1)
- Part B: LY3039478 Formulated Capsule (Test, Formulation 3) (Experimental): Single oral 50 mg dose of formulated capsule (test, formulation 3) LY3039478 administered in one of two study periods
  Interventions: Drug: LY3039478 Formulated Capsule (Test, Formulation 3)

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Part A: Placebo
Drug: LY3039478 Capsule Formulation (Formulation 3) — Administered orally
  Other Names: New Formulation
  Arms: Part A: LY3039478 Capsule Formulation (Formulation 3)
Drug: LY3039478 Drug-in Capsule (Reference, Formulation 1) — Administered orally
  Other Names: Original Formulation
  Arms: Part B: LY3039478 Drug-In Capsule (Reference, Formulation 1)
Drug: LY3039478 Formulated Capsule (Test, Formulation 3) — Administered orally
  Other Names: New Formulation
  Arms: Part B: LY3039478 Formulated Capsule (Test, Formulation 3)

SUMMARY:
The main purpose of this study is to investigate the safety of the study drug known as LY3039478 and evaluate two different formulations of LY3039478 in healthy participants. Part A has three periods. Either LY3039478 or placebo will be given once by mouth in each period. Part B has two periods. Participants will receive both formulations of LY3039478, by mouth, over the course of the study. Both parts of the study will also explore how much LY3039478 gets into the bloodstream and how long it takes the body to get rid of it. Information about any side effects will also be collected. Participants may only enroll in one part. The study will last at least 33 days, not including screening. Screening must be performed up to 30 days before enrollment.

Part B was added by protocol amendment approved in April, 2016.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m²)

Exclusion Criteria:

- Known allergies to LY3039478, related compounds or any components of the formulation

* Have previously received LY3039478
* Smokers or who have stopped smoking less than 3 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 3 treatment sequences with a placebo-control in at least 1 of the 3 study periods in Part A. Each period was separated by a washout period of ≥14 days. Participants were randomized to 1 of 2 treatment sequences in Part B. Each period was separated by a washout of ≥14 days.
Groups:
- Part A: Group 1 (25 mg LY3039478 First, Then 50 mg LY3039478, Followed by Placebo); Part A: Group 2 (25 mg LY3039478 First, Then Placebo, Followed by 75 mg LY3039478); Part A: Group 3 (Placebo First, Then 50 mg LY3039478, Followed by 75 mg LY3039478): Single oral dose of LY3039478 capsule formulation (formulation 3) administered in one of three periods.
- Part B: 50 mg LY3039478 (Reference Formulation 1 First, Then Test Formulation 3): Single oral dose of 50 mg drug-in capsule LY3039478 (reference, formulation 1) was administered in period 1, then 50 mg LY3039478 (test, formulation 3) was administered in period 2.
- Part B: 50 mg LY3039478 (Test Formulation 3 First, Then Reference Formulation 1): Single oral dose of 50 mg formulated capsule LY3039478 (test, formulation 3) administered in period 1, then 50 mg LY3039478 (reference, formulation 1) was administered in period 2.
Period: Period 1
Arm/Group | Part A: Group 1 (25 mg LY3039478 First, Then 50 mg LY3039478, Followed by Placebo) | Part A: Group 2 (25 mg LY3039478 First, Then Placebo, Followed by 75 mg LY3039478) | Part A: Group 3 (Placebo First, Then 50 mg LY3039478, Followed by 75 mg LY3039478) | Part B: 50 mg LY3039478 (Reference Formulation 1 First, Then Test Formulation 3) | Part B: 50 mg LY3039478 (Test Formulation 3 First, Then Reference Formulation 1)
Started | 5 | 5 | 5 | 7 | 7
Completed | 4 | 5 | 5 | 7 | 6
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Part A: Group 1 (25 mg LY3039478 First, Then 50 mg LY3039478, Followed by Placebo) | Part A: Group 2 (25 mg LY3039478 First, Then Placebo, Followed by 75 mg LY3039478) | Part A: Group 3 (Placebo First, Then 50 mg LY3039478, Followed by 75 mg LY3039478) | Part B: 50 mg LY3039478 (Reference Formulation 1 First, Then Test Formulation 3) | Part B: 50 mg LY3039478 (Test Formulation 3 First, Then Reference Formulation 1)
Started | 4 | 5 | 5 | 7 (Participants who completed the reference formulation in Treatment Period 1 were crossed over to receive 50 mg of the LY3039478 test formulation in Treatment Period 2.) | 6 (Participants who completed the test formulation in Treatment Period 1 were crossed over to receive 50 mg of the LY3039478 reference formulation in Treatment Period 2.)
Completed | 4 | 5 | 5 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A: Group 1 (25 mg LY3039478 First, Then 50 mg LY3039478, Followed by Placebo) | Part A: Group 2 (25 mg LY3039478 First, Then Placebo, Followed by 75 mg LY3039478) | Part A: Group 3 (Placebo First, Then 50 mg LY3039478, Followed by 75 mg LY3039478) | Part B: 50 mg LY3039478 (Reference Formulation 1 First, Then Test Formulation 3) | Part B: 50 mg LY3039478 (Test Formulation 3 First, Then Reference Formulation 1)
Started | 4 | 5 | 5 | 0 (Part B participants completed period 2 and did not participate in period 3.) | 0 (Part B participants completed period 2 and did not participate in period 3.)
Completed | 4 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in Part A and Part B.
Groups:
- Part A: Single oral dose of LY3039478 capsule formulation (formulation 3) administered in one of three periods. A washout period occurred after each period.
- Part B: Single oral dose of 50 mg drug-in capsule LY3039478 (reference, formulation 1) administered in one of two study periods. Single oral dose of 50 mg formulated capsule LY3039478 (test, formulation 3) administered in one of two study periods
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Mean Time-Matched Difference in Placebo-Adjusted QTcF Interval With Time Matched Concentrations Between LY3039478 Capsule Formulation (Formulation 3) Part A
Description: PK: mean time-matched difference in QTcF interval with time-matched concentrations between LY3039478 capsule formulation (formulation 3) compared to placebo. Analyses of QTcF was assessed by the mean change in QTcF as a function of plasma drug concentration. Triplicate measures at each time point was averaged prior to analysis. The primary analysis was based on the time-matched placebo-adjusted QTcF (ΔQTcF) for each time point, which was calculated by subtracting each participant's time-matched placebo QTcF from their QTcF results after receiving LY3039478. The relationship between plasma concentrations of LY3039478 and ΔQTcF was evaluated using a linear mixed-effects modeling approach. The response variable was ΔQTcF, and concentrations was fitted as a fixed effect with participants as a random effect. The regression slope was presented with the unit in "milliseconds per nanogram per milliliter" abbreviated as "ms/ng/mL".
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8,12, 24, 36, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable mean time-matched difference in QTcF interval data in part A. Data from all dose levels were combined due to analysis is looking at QTcF as a function of concentration of LY in the blood, not as a function of dose per protocol and statistical analysis plan.
Measure: Mean (90% Confidence Interval); unit: ms/ng/mL
Groups:
- Part A: LY3039478 Capsule Formulation (Formulation 3)+Placebo: Single oral dose of placebo, 25 mg, 50 mg, and 75 mg of LY3039478 capsule formulation (formulation 3) administered in one of three periods. A washout period occurred after each period.
Arm/Group | Part A: LY3039478 Capsule Formulation (Formulation 3)+Placebo
Number analyzed (Participants) | 15
ms/ng/mL | -0.001 [-0.006 to 0.003]

2. Secondary Outcome: PK: Cmax of LY3039478 Capsule Formulation (Formulation 3) Part A
Description: PK is Cmax of LY3039478 capsule formulation (formulation 3) in part A.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8,12, 24, 36, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 25 mg of LY3039478 capsule formulation (formulation 3 )administered in one of three periods. A washout period occurred after each period.
- Part A: 50 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 50 mg of LY3039478 capsule formulation (formulation 3) administered in one of three periods. A washout period occurred after each period.
- Part A: 75 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 75 mg of LY3039478 capsule formulation (formulation 3) or placebo administered in one of three study periods. A washout period occurred after each period.
Arm/Group | Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3) | Part A: 50 mg of LY3039478 Capsule Formulation (Formulation 3) | Part A: 75 mg of LY3039478 Capsule Formulation (Formulation 3)
Number analyzed (Participants) | 10 | 9 | 10
nanogram/milliliter (ng/mL) | 158 (43) | 296 (31) | 461 (44)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3039478 Capsule Formulation (Formulation 3) Part A
Description: PK is the area under the concentration versus time curve from zero to infinity (AUC[0-∞]) of LY3039478 capsule formulation (formulation 3) in part A.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8,12, 24, 36, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part A
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 25 mg of LY3039478 capsule formulation (formulation 3) administered in one of three periods. A washout period occurred after each period.
Arm/Group | Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3) | Part A: 50 mg of LY3039478 Capsule Formulation (Formulation 3) | Part A: 75 mg of LY3039478 Capsule Formulation (Formulation 3)
Number analyzed (Participants) | 10 | 9 | 10
nanogram*hour/milliliter (ng*h/mL) | 711 (39) | 1400 (21) | 2090 (41)

4. Secondary Outcome: PK: Cmax of the 2 Formulations of LY3039478 Part B
Description: PK is the Cmax of the 2 formulations of LY3039478 in part B
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8,12, 24, 36, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B: LY3039478 Reference, Formulation 1: Single oral dose of LY3039478 reference, formulation 1 administered in one of two study periods
- Part B: LY3039478 Test, Formulation 3: Single oral dose of LY3039478 test, formulation 3 administered in one of two study periods
Arm/Group | Part B: LY3039478 Reference, Formulation 1 | Part B: LY3039478 Test, Formulation 3
Number analyzed (Participants) | 13 | 14
ng/mL | 322 (25) | 384 (21)

5. Secondary Outcome: PK: AUC(0-∞) of the 2 Formulations of LY3039478 Part B
Description: PK is the AUC(0-∞) of the 2 formulations of LY3039478 in part B.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8,12, 24, 36, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B: LY3039478 Reference, Formulation 1 | Part B: LY3039478 Test, Formulation 3
Number analyzed (Participants) | 13 | 14
ng*h/mL | 1340 (22) | 1750 (19)

ADVERSE EVENTS:
Groups:
- Part A: Placebo: Single oral dose placebo administered in one of three study periods. A washout period occurred after each period.
- Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 25 mg of LY3039478 capsule formulation (formulation 3) administered in one of three periods.
- Part A: 50 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 50 mg of LY3039478 capsule formulation (formulation 3) administered in one of three periods.
- Part A: 75 mg of LY3039478 Capsule Formulation (Formulation 3): Single oral dose of 75 mg of LY3039478 (formulation 3) or placebo administered one of three study periods.
Arm/Group | Part A: Placebo | Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3) | Part A: 50 mg of LY3039478 Capsule Formulation (Formulation 3) | Part A: 75 mg of LY3039478 Capsule Formulation (Formulation 3) | Part B: LY3039478 Reference, Formulation 1 | Part B: LY3039478 Test, Formulation 3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/9 | 0/10 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/10 | 1/9 | 0/10 | 1/13 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=14) | Part A: 25 mg of LY3039478 Capsule Formulation (Formulation 3) (N=10) | Part A: 50 mg of LY3039478 Capsule Formulation (Formulation 3) (N=9) | Part A: 75 mg of LY3039478 Capsule Formulation (Formulation 3) (N=10) | Part B: LY3039478 Reference, Formulation 1 (N=13) | Part B: LY3039478 Test, Formulation 3 (N=14)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days